CLINICAL TRIAL: NCT02103634
Title: NaF PET/MRI Evaluation for Bone Metastases in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE5113
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Malignant Neoplasm of Breast TNM Staging Distant Metastasis (M); Untreated Bone Metastases
Keywords: breast cancer; FDG PET/CT; MRI; NaF PET/MRI; NaF PET/CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Lesion Imaging: Image patients with the standard of care of a FDG PET/CT and the experimental method of the NaF PET/MRI and compare the number of images found within and between patients to determine the most effective way of looking at breast cancers metastasized to bone
  Interventions: Device: NaF PET/MRI; Device: NaF PET/CT; Device: FDG PET/CT

INTERVENTIONS:
Device: NaF PET/MRI
Device: NaF PET/CT — NaF PET/CT images will be obtained through fusion software. Researchers will fuse the Non AC and AC NaF images with the low dose CT obtained in the FDG PET/CT study.
Device: FDG PET/CT

SUMMARY:
This study will look at two new technologies being developed for measuring cancer in bones. One of these technologies is a substance called Sodium Fluoride (NaF). Fluoride is a normal body substance. The amount that patients will receive has been shown to be very safe. One study of over 400 patients showed no adverse reactions after receiving the recommended dosage.

NaF (known as a radiotracer) is taken up into the bones under a normal process and researchers can measure the amount within patient's bones through an imaging system called a Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI). This system combines aspects of both a PET study as part of the regular standard of care and an MRI study. The belief is that the combination of these two studies will be better than either study alone.People who have enrolled in this study will receive their clinically requested PET/CT scan as part of their normal diagnostic care and will follow all the said recommendations for this study such as not being pregnant, having fasted overnight, etc. Subjects will return within 7 days for a 10 mCi NaF PET/MRI study. The patients' imaging time will be up to 120 minutes depending on the MRI sequences acquired. Imaging for the PET portion of the study will take approximately 20-30 minutes with the rest of the time devoted to MRI sequences.

DETAILED DESCRIPTION:
The primary aim of this study is to assess NaF PET/MRI compared to NaF PET/CT and standard of care imaging made available for assessment of bone metastases in all cancers as well as other standard of care indications for MDP bone scintigraphy. The study will use both the currently available and approved MRI sequences for attenuation correction and localization as well as non FDA approved sequences to assess the ability of the modality to identify bone metastases.

Study Goals:

1. Assess the sensitivity, specificity, accuracy of NaF PET/MRI vs. Naf PET/CT vs. current standard of care imaging. This will be done on a lesion by lesion basis based on a prior study looking at NaF PET/CT (14). Lesions that are positive on NaF PET/MRI but not on other imaging will be followed up on future imaging to see if they eventually become positive given that physiology changes before anatomy. Follow up will include both repeat NaF PET/CT (PET/MRI) studies (as per standard of care MDP bone scintigraphy indications) as well as review of other surveillance standard of care imaging up to 6 months after the NaF PET/CT (PET/MRI) was done.
2. Assess various NaF MRI sequences for attenuation correction and localization both from approved and developmental sequences compared to NaF CT attenuation corrected images through software.
3. Assess the ability of MRI sequences acquired for attenuation correction and localization to evaluate bone metastases in comparison to other modalities.
4. Assess the image quality of various NaF MRI sequences acquired for attenuation correction and localization using both approved and developmental sequences.
5. Ascertain, if there are lesions identified on the NaF PET/MRI study but not seen on the NaF PET/CT study (or other standard of care imaging) or vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Referred to University Hospitals Cleveland Medical Center Nuclear Medicine for methylene diphosphonate (MDP) Bone Scintigraphy
* Must understand and voluntarily sign an Informed consent form after the contents have been fully explained to them.
* Patients must have no contra-indications to PET/CT or MRI (Patients will NOT be receiving either CT or MRI contrast and thus, those contraindications are not exclusionary).

Exclusion Criteria:

* Patients who cannot tolerate imaging up to 120 minutes of total imaging (breaks of several minutes between imaging will be available)
* Pregnant or breast feeding women.
* Healthy volunteers
* Inability to comply with instructions
* MRI contraindications Include:

  * Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips
  * Patients with implanted pacemaker or implanted defibrillator device
  * Patients with contraindications for MRI due to embedded foreign metallic objects. Bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient
  * Implanted medical device not described above that is not MRI-compatible
  * Known history of claustrophobia
  * Contrast contraindications not included since patients will not be receiving MRI or CT contrast as part of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who present for bone imaging as per Tc-methylene diphosphonate (MDP) bone scan standard of care indications
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity of NaF PET/MRI | 2 years after beginning of study
  The difference in the number of lesions detected by the two imaging methods using McNamar's test

SECONDARY OUTCOMES:
Image Quality | 2 years after beginning of study
  Mean quality score ranging from 1-5 using different methods will be compared using paired t-tests. With a sample size of 150 lesions, a difference of 0.25 points in mean quality score can be detected with 86% power.
Positive predictive value of MRI sequences | 2 years from beginning of study
  The difference in positive predictive value of bone metastases detected by MRI sequences as compared to other modalities as calculated using McNamar's test.
Negative predictive value of MRI sequences | 2 years from beginning of study
  The difference in Negative predictive value of bone metastases detected by MRI sequences as compared to other modalities as calculated using McNamar's test.
Specificity of MRI sequences | 2 years from beginning of study
  The difference in specificity of bone metastases detected by MRI sequences as compared to other modalities as calculated using McNamar's test.
attenuation correction | 2 years after beginning of study
  Difference in attenuation correction of NaF MRI-based and NaF CT-based images as calculated using McNamar's test.
localization | 2 years after beginning of study
  Difference in localization of NaF MRI-based and NaF CT-based images as calculated using McNamar's test.
Evaluation of Bone Metastases | 2 years after beginning of study
  Difference in bone metastases detected by MRI attenuation correction images compared to diagnostic quality images.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Jones, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States